CLINICAL TRIAL: NCT02072928
Title: Study of Botulinum Toxin Type A (BOTOX®) to Treat Urinary Incontinence From Neurogenic Detrusor Overactivity in Belgium
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/NS/OAB/005
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- BOTOX®: Patients with incontinence from NDO due to spinal injury or MS prescribed BOTOX® (Botulinum toxin Type A) as standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A (BOTOX®) prescribed as standard of care in clinical practice.
  Other Names: onabotulinumtoxinA; BOTOX®

SUMMARY:
This study will evaluate the impact of BOTOX® treatment on anticholinergic drug use in patients with urinary incontinence from Neurogenic Detrusor Overactivity (NDO) due to spinal injury or Multiple Sclerosis (MS) who are prescribed BOTOX® as standard of care in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed BOTOX® for urine incontinence from NDO due to spinal injury or MS as standard of care in clinical practice in Belgium
* Previous treatment with anticholinergic drugs ineffective
* Last BOTOX® treatment ≥18 months.

Exclusion Criteria:

* Diagnosis of urinary incontinence less than 9 months.
* No anticholinergic drug use in the last 9 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with incontinence from NDO due to spinal injury or MS treated as per standard of care in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-01-28 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2015-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (6):
- Belgium (6):
  - UZA, Edegem
  - CHU de Liège, Esneux
  - UZ Gent, Ghent
  - Centre Hospitalier Regional de Huy, Huy
  - UZ Leuven, Leuven
  - Maria Ziekenhuis Noord-Limburg, Overpelt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BOTOX®
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BOTOX®
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Anticholinergic Drug Use
Description: Anticholinergic drug use was collected the 9 months before the baseline Botox® treatment and the 9 months following the baseline Botox® treatment. Total anticholinergic drug use in the 9 months following the baseline Botox® treatment is noted.
Time Frame: Baseline, 9 Months
Population: Treatment responders for whom pharmacy data is available
Measure: Mean (Standard Error); unit: Doses of Anticholinergic Drugs
Arm/Group | BOTOX®
Number analyzed (Participants) | 47
Doses of Anticholinergic Drugs
  Baseline | 305.21 (36.94)
  9 Months | 199.77 (40.46)

ADVERSE EVENTS:
Description: All enrolled patients were used to assess adverse events and serious adverse events.
Arm/Group | BOTOX®
Serious Adverse Events (participants affected / at risk) | 4/55
Other Adverse Events (participants affected / at risk) | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | BOTOX® (N=55)
Epididymitis (Reproductive system and breast disorders) | 1/28
Pyelonephritis (Renal and urinary disorders) | 1
Progression of MS (Respiratory, thoracic and mediastinal disorders) | 1
Erysipelas (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.